CLINICAL TRIAL: NCT04788706
Title: Efficacy of Low-level Laser Therapy Associated With Russian Electrical Stimulation in Knee Osteoarthritis: a Randomized Controlled Double-blind Study
Brief Title: LLLT and Russian Electrical Stimulation in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0775/08
Record Dates: First submitted 2020-12-29; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2020-12

CONDITIONS: Osteo Arthritis Knee
Keywords: low level laser therapy; Russian electrical stimulation
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Active Comparator): LLLT over three weeks followed by an eight-week receiving Russian electrical stimulation
  Interventions: Other: Low level Laser Therapy and Russian electrical stimulation
- Group II (Placebo Comparator): Placebo laser over three weeks followed by an eight-week receiving Russian electrical stimulation
  Interventions: Other: Placebo Laser and Russian electrical stimulation
- Group III (Active Comparator): LLLT over three weeks followed by an eight-week receiving LLLT application combined with Russian electrical stimulation
  Interventions: Other: Low level Laser Therapy and Low level Laser Therapy plus Russian electrical stimulation
- Group IV (Placebo Comparator): Placebo laser over three weeks followed by an eight-week receiving Placebo laser application combined with Russian electrical stimulation
  Interventions: Other: Placebo Laser and Placebo Laser plus Russian electrical stimulation

INTERVENTIONS:
Other: Low level Laser Therapy and Russian electrical stimulation — LLLT over three weeks followed by an eight-week receiving Russian electrical stimulation
  Arms: Group I
Other: Placebo Laser and Russian electrical stimulation — Placebo laser over three weeks followed by an eight-week receiving Russian electrical stimulation
  Arms: Group II
Other: Low level Laser Therapy and Low level Laser Therapy plus Russian electrical stimulation — LLLT over three weeks followed by an eight-week receiving LLLT application combined with Russian electrical stimulation
  Arms: Group III
Other: Placebo Laser and Placebo Laser plus Russian electrical stimulation — Placebo laser over three weeks followed by an eight-week receiving Placebo laser application combined with Russian electrical stimulation
  Arms: Group IV

SUMMARY:
Objectives: To investigate the effect of low-level laser therapy (LLLT) application combined with Russian Electrical Stimulation on pain, mobility, functionality, range of motion, muscular strength, and activity in patients with osteoarthritis of the knee.

Design: Randomized controlled double-blind study. Setting: Specialist Rehabilitation Services.

DETAILED DESCRIPTION:
ABSTRACT Objectives: To investigate the effect of low-level laser therapy (LLLT) application combined with Russian Electrical Stimulation on pain, mobility, functionality, range of motion, muscular strength, and activity in patients with osteoarthritis of the knee.

Design: Randomized controlled double-blind study. Setting: Specialist Rehabilitation Services. Participants: Eighty participants with knee osteoarthritis were randomized. Intervention: Participants were randomized into four groups: Group I (n=20; LLLT over three weeks followed by an eight-week receiving Russian electrical stimulation), Group II (n=20; Placebo laser over three weeks followed by an eight-week receiving Russian electrical stimulation), Group III (n=20; LLLT over three weeks followed by an eight-week receiving LLLT application combined with Russian electrical stimulation), Group IV (n=20; Placebo laser over three weeks followed by an eight-week receiving Placebo laser application combined with Russian electrical stimulation). The groups treated with LLLT received treatments with invisible infrared laser (904 nm, 3 Joules/point). The Placebo groups received identical treatment, but the infrared laser output was disabled. The sessions occurred three times a week.

Main outcome measures: The primary outcome was the change in knee pain and functionality (Lequesne). Secondary outcomes included change in mobility (8 meters and Timed Up and Go test), range of motion (goniometer), muscular strength (dynamometer), activity (Western Ontario and McMaster Universities Osteoarthritis questionnaire) and medication intake.

ELIGIBILITY:
Inclusion Criteria:

1. levels 2-4 according to Kellgren-Lawrence grade
2. aged 50-75 years
3. both genders
4. have knee pain and functional disability for at least three months
5. according to the criteria of the American College for Rheumatology.

Exclusion Criteria:

* cancer, diabetes, symptomatic hip osteoarthritis, or used antidepressants, anti-inflammatory medications or anxiolytics during six months prior to enrolment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 6 months from baseline (follow up)
  numeric pain rating scale (0-10) with a minimal clinically important change of two points
Functionality | 6 months from baseline (follow up)
  Was measured using the Lequesne questionnaire (11 questions about pain, discomfort and function). Scores range from 0 to 24 (from 'no' to 'extremely severe' dysfunction).

SECONDARY OUTCOMES:
Medication intake | 6 months from baseline (follow up)
  Paracetamol
Mobility and balance | 6 months from baseline (follow up)
  were evaluated by the Timed Up and Go (TUG) test19 and the 8-meter walk test.20 The TUG test, a measure of functional mobility, quantifies in seconds the time that the individual needs to stand up from a chair, walk 3m, turn back toward the chair and sit down again. The 8-meter walk test measures the time and number of steps required for a person to walk 8m.
Range of motion of the knees | 6 months from baseline (follow up)
  was measured with a universal goniometer (AESCULAP).
Muscular strength | 6 months from baseline (follow up)
  was estimated at maximal isometric force for the quadriceps, using a portable dynamometer (Lafayette, USA). Under stabilized conditions, patients, sitting with knees flexed at 60 (measured by a goniometer),21 were asked to extend the legs as far as they could. Three trials were conducted, and the mean value was obtained.
Activity | 6 months from baseline (follow up)
  was measured using the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) questionnaire,22 which is self-administered and measures pain, frozen joints and physical activity. Increased scores suggest decreased activity.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia P Alfredo, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Department of Physical Therapy, Speech and Occupational Therapy of University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The results obtained with the study will be made available to participants at the end of the study. These data will be published in articles, so that the anonymity of the participants is guaranteed.
  All subjects who agreed to participate in the study signed a free and informed consent form and authorized the dissemination of the study results in articles or abstracts presented at scientific congresses.